CLINICAL TRIAL: NCT05875623
Title: Impact of Medications Review on Potentially Inappropriate Medications and Clinical Outcomes Among Hospitalized Older Adults: A Randomized Controlled Trial (REVMED RCT) Protocol
Brief Title: Impact of Medications Review on Potentially Inappropriate Medications and Clinical Outcomes Among Hospitalized Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Hospital Raja Permaisuri Bainun (Other Government)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REVMED RCT
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-11

CONDITIONS: Deprescriptions; Aged; Inappropriate Prescribing; Potentially Inappropriate Medications; Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In the intervention group, the clinical pharmacist will apply the MALPIP criteria on all the admission and discharge medications. The pharmacists can access the full MALPIP list at https://sites.google.com/moh.gov.my/malpip/home.
  The intervention will consist of 4 steps: i) pharmacist review using MALPIP criteria to detect PIM, ii) discussion with doctors for deprescribing decision iii) discussion with patients and documentation of shared decision iv) follow up patients at 6, 12, and 18 months.
  Pharmacists will perform the reviewing and checking by themselves and discuss the suggestions with doctors during daily medical ward rounds. The attending doctors will decide whether to deprescribe based-on pharmacists suggestions. Then, the pharmacists will discuss the deprescribing proposal with the patients and record the decision.
  Interventions: Other: MALPIP criteria
- Control (No Intervention): In the control arm, pharmacists, patients and doctors are not purposefully blinded but are not aware of the intervention (i.e. the MALPIP tool). Designated pharmacist at the control sites identifies patients who match the eligibility requirements and enroll them into the trial after obtaining consent.
  Patients in the control arm will receive routine care and support that they entitled to from the medical team and clinical pharmacists. Preadmission medication will be reconciled by a clinical pharmacist using the standard procedures, including medication history assessment form (CP1), pharmacotherapy review (CP2) and the clinical pharmacy report form (CP3).

INTERVENTIONS:
Other: MALPIP criteria — In the intervention group, the clinical pharmacist will apply the MALPIP criteria on all the admission and discharge medications. The intervention will consist of 4 steps: i) pharmacist review using MALPIP criteria to detect PIM, ii) discussion with doctors for deprescribing decision iii) discussion with patients and documentation of shared decision iv) follow up patients
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to assess the effectiveness of a pharmacist-led medication review using the locally developed Malaysian Potentially Inappropriate Prescribing Screening tool in Older Adults (MALPIP), an explicit criteria in hospitalized older adults. The main questions it aims to answer are:

1. The effectiveness of the intervention in reducing the number of PIMs and chronic medications after discharge
2. The impact of the intervention on quality of life, falls events, emergency department visits, readmissions and survivals

Researchers will compare the control group to see if there is corresponding changes to the outcomes specified above.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years and above
* Taking more than five regular drugs
* Having at least one chronic medical condition
* Ability to understand and speak Malay, English, or Mandarin language

Exclusion Criteria:

* Admitted for end-of-life care
* Diagnosed with terminal illness
* Diagnosed with active cancer
* Participated in another drug trial
* Refused or unable to give consent
* Visited the Emergency Department without admission to ward
* Readmitted and have been previously enrolled in the trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of potentially inappropriate medications | Admission up to 18 months
Number of chronic medications | Admission up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Chee Tao Chang, Msc, Principal Investigator — Monash University Malaysia
Locations (1):
- Shaun Lee, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang CT, Teoh SL, Cheah WK, Lee PJ, Azman MA, Ling SH, Chuah ASC, Sabki NH, George D, Oh HL, Goh JY, Lee SH, Foong WK, Lee JCY, Chan HK, Teoh LR, Lim XJ, Rajan P, Lee SWH. Impact of deprescribing intervention on potentially inappropriate medications and clinical outcomes among hospitalized older adults in Malaysia: a randomized controlled trial (REVMED RCT) protocol. J Pharm Policy Pract. 2023 Oct 3;16(1):113. doi: 10.1186/s40545-023-00621-5. PMID 37789376